CLINICAL TRIAL: NCT01841463
Title: An Open Label, Multicenter, Phase I Extension Study of an Oral Cdk Inhibitor P1446A-05 Administered With an Oral BRAF Inhibitor Vemurafenib (Zelboraf®) in Patients With Advanced or Inoperable Malignant Melanoma With BRAF Mutation
Brief Title: Study of an Oral Cdk Inhibitor Administered With an Oral BRAF Inhibitor in Patients With Advanced or Inoperable Malignant Melanoma With BRAF Mutation
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision not related to patient safety
Sponsor: Piramal Enterprises Limited (Industry)
Collaborators: Melanoma Research Foundation Breakthrough Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1446A-05/72/12
Record Dates: First submitted 2013-04-17; First posted 2013-04-26 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Advanced or Inoperable Malignant Melanoma With BRAF Mutation
Keywords: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P1446A-05 (Experimental): * The study will be conducted in two phases- Phase I ('Dose escalation' phase), and Extension phase:-
  * In the 'Dose escalation' phase patients will be co-administered P1446A-05 (150, 250, 350 mg qd) and vemurafenib (720, 960 mg bid) in a cohort of three to six patients on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity.
  * In the 'Extension' phase, sixty patients with BRAF V600E/K mutations (forty patients naïve to selective BRAF inhibitor therapy, and twenty progressing on selective BRAF inhibitor therapy) will be treated at the MTD on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity
  Interventions: Drug: P1446A-05; Drug: Vemurafenib (Zelboraf®)

INTERVENTIONS:
Drug: P1446A-05 — - In the 'Dose escalation' phase patients will be co-administered P1446A-05 (150, 250, 350 mg qd) & vemurafenib (720, 960 mg bid) in a cohort of 3 to 6 patients on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity. The next higher dose during the dose escalation phase will depend upon demonstrated safety in the previous dose group. The max tolerated dose (MTD) of P1446A-05 & vemurafenib co-administered will be determined. In the 'Extension' phase, 60 patients with BRAF V600E/K mutations (40 patients naïve to selective BRAF inhibitor therapy, & 20 progressing on selective BRAF inhibitor therapy) will be treated at the MTD on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity to determine efficacy of the co-administration. Additionally, there will be a cohort of 10 patients who consent for mandatory serial tumor biopsy samples & undergo 'Monotherapy' for 14 days with P1446A-05 at the MTD of the co-administration.
Drug: Vemurafenib (Zelboraf®) — * In the 'Dose escalation' phase patients will be co-administered P1446A-05 (150, 250, 350 mg qd) and vemurafenib (720, 960 mg bid) in a cohort of 3 to 6 patients on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity. Escalation to the next higher dose during the dose escalation phase will depend upon demonstrated safety in the previous dose group. The maximum tolerated dose (MTD) of P1446A-05 and vemurafenib co-administered will be determined.
  * In the 'Extension' phase, 60 patients with BRAF V600E/K mutations (40 patients naïve to selective BRAF inhibitor therapy, and 20 progressing on selective BRAF inhibitor therapy) will be treated at the MTD on a 28-day cycle
  * Additionally, there will be a cohort of 10 patients who consent for mandatory serial tumor biopsy samples and undergo 'Monotherapy' for 14 days with P1446A-05 at the MTD of the co-administration.

SUMMARY:
* An Open Label, Multicenter, Phase I Extension Study of an Oral Cdk Inhibitor P1446A-05 Administered with an Oral BRAF Inhibitor Vemurafenib (Zelboraf®) in Patients with Advanced or Inoperable Malignant Melanoma with BRAF Mutation
* The primary objective is to determine the safety, maximum tolerated dose (MTD), and dose limiting toxicity (DLT) of the co-administration of P1446A-05 with vemurafenib, in melanoma patients with BRAF mutation

ELIGIBILITY:
Inclusion Criteria:

1. Patients having histologically confirmed unresectable (Stage III) or metastatic (Stage IV) malignant melanoma with a positive BRAF mutation result determined by Roche CoDx or local CLIA-certified analysis
2. Patients naïve to a selective BRAF inhibitor therapy or must have progressed after therapy on a selective BRAF inhibitor. For patients entering the protocol progressing on vemurafenib therapy, they must be tolerant of the 960 mg po bid dose.
3. Tumor biopsies are optional in this study except for patients entering the mandatory biopsy cohorts. Nevertheless tumor biopsies are encouraged, especially in patients with accessible tumors for biopsy to include the collection of formalin-fixed, paraffin-embedded (FFPE) and fresh- frozen tissue (FF) as outlined in the biomarker sections of the protocol. Willingness of patient to give consent of biopsy, should be ascertained
4. Patients of ≥ 18 years of age
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0 or1
6. Patients with measurable disease per 'Response Evaluation Criteria In Solid Tumors' (RECIST version 1.1)
7. Patients must have normal organ and adequate marrow function
8. Patients with ability to swallow and retain oral medication
9. Women of childbearing potential and men willing to agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilized.
10. Negative serum pregnancy test within 10 days prior to commencement of therapy dosing in premenopausal women. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year.
11. Ability to understand and the willingness to offer a written Informed Consent document prior to the screening procedures for participation into the study

    * For Extension phase-
    * For patients entering the protocol progressing on vemurafenib therapy, they must be tolerant of the vemurafenib dose selected for the extension phase

Exclusion Criteria:

1. Prior malignancy (within the last 2 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or any other cancer for which the patient has been disease-free for at least 2 years
2. Patients who have received any prior chemotherapy, radiotherapy, biologic/targeted anti-cancer therapy (one week for BRAF inhibitor for melanoma) or surgery within 4 weeks (6 weeks for monoclonal antibodies, radioactive monoclonal antibodies or any radio-or toxin-immunoconjugates) before Day 1 of Investigational product administration and have not recovered (to < Grade 1) from the toxic effects from any prior therapy
3. Patients having received any other investigational agents within 4 weeks prior to Day 1 of Investigational product administration and have not recovered completely (to < Grade 1) from the side effects of the earlier investigational agent
4. Anticipated administration of any anti-cancer therapies (chemotherapy, radiation therapy, immunotherapy, biological therapy, hormonal therapy, surgery, and/or tumor embolisation) other than those administered in this study such as BRAF inhibitor
5. Patients with symptomatic or untreated leptomeningeal or brain metastases, or spinal cord compression [patients with previous brain metastases will be allowed to enter the trial if metastases have been surgically removed or all known sites of metastases have been treated with stereotactic high dose radiosurgery. Patients must be off corticosteroids for at least one month and have a stable lesion with verification by imaging (CT/MRI) within 28 days prior to Day 1 of Investigational product administration]
6. Patients with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic diarrheal condition, refractory nausea, vomiting or any other condition that will interfere significantly with the absorption of study drugs
7. Patients with mean QTc interval >480 msec at screening
8. Treatment with drugs with potential to cause dysrhythmias including but not limited to terfenadine, quinidine, procainamide, diisopyramide, sotalol, probucol, bepridil, haloperidol, risperidone and/or indapamide
9. Patients on warfarin treatment
10. Any condition for which participation in this study as judged by the Investigator to be detrimental to the patient with (such as) inter-current illness including, but not limited to ongoing or active infection, New York Heart Association functional classification class III, or IV heart failure; unstable angina pectoris; cardiac arrhythmia; history of myocardial infarction; uncontrolled hypertension (blood pressure above 160/100 mm Hg despite antihypertensive treatment); coronary artery bypass graft; cerebrovascular accident; transient ischemic attack or pulmonary embolism during the previous 6 months or psychiatric illness/social situations that would jeopardize compliance with study requirements
11. Patients with a known immediate or delayed hypersensitivity reaction or idiosyncrasy to any other medication chemically related to P1446A-05 or vemurafenib, or excipients considered to be clinically significant by the investigator
12. Nursing woman
13. Patients with known HIV positivity or AIDS- related illness, or active Hepatitis B virus, and active Hepatitis C virus
14. Patients taking drugs known to prolong the QTc interval who cannot be switched to an alternative drug.

For Extension phase-

1. Patients with active second malignancy will be eligible as long as they do not need systemic therapy for the second malignancy
2. Patients with active brain metastases will be included in the study as long as the tumor size is less than 1 cm without the requirement of steroid use for neurological symptoms
3. Patients with evaluable metastatic disease will be allowed even if there is no measurable disease per RECIST 1.1. In this case patients with many sub centimeter in-transit skin/SQ nodules will be eligible for the biopsy cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Dose Limiting Toxicity | Until disease progression or unacceptable toxicity (expected to be 6-8 months)
  The study will be conducted in two phases- Phase I (Dose escalation phase), and Extension phase. In the Dose escalation' phase patients will be co-administered P1446A-05 (150, 250, 350 mg qd) and vemurafenib (720, 960 mg bid) in a cohort of three to six patients on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity. Escalation to the next higher dose during the dose escalation phase will depend upon demonstrated safety in the previous dose group. The maximum tolerated dose (MTD) of P1446A-05 and vemurafenib co-administered will be determined. In the 'Extension' phase, sixty patients with BRAF V600E/K mutations (forty patients naïve to selective BRAF inhibitor therapy, and twenty progressing on selective BRAF inhibitor therapy) will be treated at the MTD on a 28-day cycle, until the occurrence of disease progression or unacceptable toxicity to determine efficacy of the co-administration.

SECONDARY OUTCOMES:
Tumor Response | Until disease progression or unacceptable toxicity (expected to be 6-8 months)
  - To determine best Overall Response Rate (ORR), Duration of response (DOR), Progression Free Survival (PFS), and Overall Survival (OS) of the co-administration of P1446A 05 and vemurafenib using RECIST version 1.1 in melanoma patients with BRAF mutation
Pharmacokinetic (PK) | Cycle1 (Day 15 and 22) and Cycle 2 (Day1,15 and 28)
  * PK parameters such as Cmax, Tmax, AUC0-t, AUC0-inf, Kel, CL, Vz and t1/2 will be determined using standard non-compartmental and population pharmacokinetic approach (wherever possible).
  * Blood samples (6 mL at each time point) for pharmacokinetic assessment will be collected at the following time points in Dose Escalation Phase- Cycle 1- Day 15: pre-dose (within 30 min before swallowing the capsule/s, 1, 2, 4, 6, 8hr; Day 19: pre-dose (within 30 min before swallowing the capsule/s, 1, 2, 4, 8hr; and within one hour post dose on Day 22.
  * Additionally, blood samples for PK analysis may be collected should patient develop SAE at the earliest feasible time point.
Biomarker Analysis | Until disease progression or unacceptable toxicity (expected to be 6-8 months)
  * The biomarkers will be assessed pre- and post-treatment and will focus on (a) inhibition of the MAPK pathway as a target of vemurafenib, a RAF inhibitor; (b) cell cycle pathways as an effect of P1446A-05, a Cdk inhibitor; (c) mechanisms of resistance; and (d) markers for senescence and apoptosis as evidence of target engagement/drug response.
  * During phase I dose escalation, optional tumor samples will be collected at screening, within 4 to 6 hours of drug administration on Day 14 of Monotherapy and between Cycle 1 Day 15 and Cycle 1 Day 21, and at disease progression
  * After the MTD is determined, 10 additional patients will be enrolled in "Serial Tumor biopsy cohort"
  * During the Extension phase, tumor samples will be collected at screening, Cycle 1 Day 15 and Cycle 1 Day 21 within 4 to 6 hours of drug administration, and at disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, MD, Principal Investigator — UCSF Medical Center at Mount Zion; Kevin B Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - UCSF Medical Center at Mount Zion, South San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Georgetown-Lombardi Comprehensive Cancer Ctr, Washington D.C., District of Columbia
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas